CLINICAL TRIAL: NCT00448942
Title: The Impact of the Use of Chlorhexidine-Based Bathing System in the Hospital to Reduce the Incidence of MRSA/VRE Infection or Colonization and Nosocomial Bloodstream Infections (BSI)
Brief Title: The Impact of Chlorhexidine-Based Bathing on Nosocomial Infections
Status: Completed | Type: Observational
Sponsor: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Collaborators: Weill Medical College of Cornell University (Other); Washington University School of Medicine (Other); Johns Hopkins University (Other); University of Tennessee (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Other Study IDs: 01115; UR8/CCU315346-03-1
Record Dates: First submitted 2007-03-15; First posted 2007-03-19 (Estimated); Last update posted 2007-03-19 (Estimated); Status verified 2007-03

CONDITIONS: Nosocomial Bacteremia; Nosocomial Fungemia; MRSA Colonization; MRSA Infection; VRE Colonization; VRE Infection
Keywords: Staphylococcus aureus [B03.510.400.790.750.100]; Enterococcus faecalis [B03.510.400.800.280.280]; Enterococcus faecium [B03.510.400.800.280.300]; Bacteremia [C01.252.100]; Fungemia [C01.703.360]; Infection Control [G03.850.780.200.450]; Antisepsis [G03.850.780.200.450.150]

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Daily bathing with Chlorhexidine based product

SUMMARY:
The purpose of this study was to determine if the use of daily chlorhexidine bathing would decrease the incidence of MRSA and VRE colonization and healthcare associated Bloodstream Infections (BSI) among Intensive Care Unit (ICU) patients.

DETAILED DESCRIPTION:
Infections due to Staphylococci including MRSA are the predominant nosocomially acquired complication in the intensive care unit. The increasing incidence of MRSA colonization and infection among ICU patients has been attributed to many factors including increased admission of patients already colonized with MRSA to the ICU, poor compliance with handwashing and barrier precautions, delayed identification of MRSA colonized patients, and understaffing. Measures that have proven to limit horizontal transmission between patients and staff and staff to patients include strict attention to barrier precautions and handwashing. Unfortunately both of these strategies require levels of compliance that are often not achieved.

Nosocomial blood stream infections are a leading source of morbidity and mortality among intensive care unit patients. Several modifiable factors have been shown to increase the risk of bloodstream infections. These include lapses in the use of strict sterile technique in the insertion of central venous catheters and improper site preparation. New CDC guidelines on the prevention of catheter related bloodstream infections recommend that the preferential use of chlorhexidine containing skin disinfectants be used for site preparation prior to insertion. The use of chlorhexidine reduces residual skin organisms as well as inhibits their rebound growth and has been demonstrated to reduce catheter-associated bloodstream infections in comparison to other skin disinfectant products such as povidone-iodine.

As a result of guidelines promoting the use of chlorhexidine, a number of intensive care units have implemented quality improvement projects examining the potential role of chlorhexidine based bathing of intensive care unit patients in reducing nosocomial transmission of multiresisitant organisms such as MRSA and vancomycin-resistant enterocooci (VRE). The goal of the currently proposed study is to analyse existing data from participating intensive care units that have adopted the use of chlorhexidine antisepsis to determine the impact of chlorhexidine on bacterial colonization and nosocomial infections Participating hospitals who have completed quality improvement projects that included the use of chlorhexidine in bathing of ICU patients will submit de-identified data on nosocomial bacteremias and MRSA and VRE colonization during defined time periods where chlorhexidine bathing was used in comparison to time periods where regular bathing procedures were utilized.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients admitted to study units

Exclusion Criteria:

* Children under the age of 18
* Previous adverse reaction or documented allergy to chlorhexidine based products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5300
Dates: Start 2004-11; Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward W Wong, MD, Principal Investigator — Hunter Holmes Mcguire Veteran Affairs Medical Center
Locations (4):
- United States (4):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Barnes Jewish Hospital, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Hunter Holmes McGuire Veteran Affairs Medical Center, Richmond, Virginia